CLINICAL TRIAL: NCT01203735
Title: Valproic Acid in Combination With Concurrent Chemoradiotherapy Using Vinorelbine and Cisplatin for Inoperable Locally Advanced Non-Small-Cell Lung Cancer
Brief Title: Valproic Acid With Chemoradiotherapy for Non-Small-Cell Lung Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Dr. Konstantin Lavrenkov, MD, PhD, Department of Oncology, Soroka University Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOR507910CTIL
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2011-03-29 (Estimated); Status verified 2010-09

CONDITIONS: Locally Advanced Inoperable Non-small-lung Cancer
Keywords: Non-small-cell lung cancer; Valproic acid; Chemotherapy; Radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Valproic acid, Chemoradiotherapy (Other)
  Interventions: Drug: Valproic acid

INTERVENTIONS:
Drug: Valproic acid — 800mg per day for entire period of RT
  Other Names: Sodium valproate

SUMMARY:
This is non-randomized phase 2 study to evaluate toxicity and efficacy of VA with concurrent chemoradiotherapy (CCRT) containing weekly vinorelbine and cisplatin in patients with locally advanced inoperable non-small-cell lung cancer (NSCLC).All patients will be planned for three-dimensional conformal RT (3-DCRT). Concurrent weekly vinorelbine and cisplatin and oral valproic acid (VA)will be started at the first day of RT. Follow up will be conducted every 3 months after completion of the study treatment. Toxicity will be assessed using CTCAE, based on clinical examination and laboratory tests during the study treatment and at follow up visits. Response to treatment will be evaluated using RECIST criteria. Overall and progression free survival (OS and PFS) will be estimated using the Kaplan-Meier method.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years.
2. Newly-diagnosed, histologically or cytologically confirmed NSCLC.
3. Inoperable stage IIIA-B disease
4. KPS > 60
5. FEV1 >1.2L
6. No previous RT to chest
7. No serious comorbid condition
8. No treatment with biological response modifiers or cytotoxic agents within four weeks prior to study entry
9. No participation in clinical trial using any investigational drug or device within four weeks prior to study entry
10. No serious complication of malignant condition
11. No previous or concurrent malignancy at other sites except cone biopsied in situ carcinoma of the uterine cervix and adequately treated basal cell or squamous cell carcinoma of the skin
12. Adequate organ function as evidenced by the following peripheral blood counts or serum chemistries at study entry:

    Hemoglobin > 9.0 Gm/dL WBC count > 4.0x109/L Neutrophile count > 1.5 cells x 109/L, Version 1, May 12, 2010 Platelet count > 100 x 109/L, Creatinine < 1.5 mg/dL Total bilirubin < upper limit of normal (ULN) AST/SGOT < ULN Calcium < ULN
13. Ability to sign informed consent
14. Ability to attend follow-up visits

Exclusion Criteria:

1. Operable disease
2. Metastases to contra-lateral mediastinal lymph nodes
3. Distant metastases
4. KPS < 60
5. FEV1 < 1.2L
6. Previous RT to chest
7. Treatment with biological response modifiers or cytotoxic agents within four weeks prior to study entry
8. Participation in clinical trial using any investigational drug or device within four weeks prior to study entry
9. Major surgical procedure within two weeks prior to study entry
10. Serious comorbid condition, inclusive but not limited to myocardial infarction within previous six months, uncontrolled cardiac arrhythmias, uncontrolled angina pectoris, active infection including acute hepatitis
11. Serious complication of malignant condition
12. Previous or concurrent malignancy
13. Inadequate organ function as evidenced by the following peripheral blood counts or serum chemistries at study entry:

    Hemoglobin < 9.0 Gm/dL WBC count < 4.0x109/L Neutrophile count < 1.5 cells x 109/L, Platelet count < 100 x 109/L, Creatinine > 1.5 mg/dL Total bilirubin > ULN (upper limit of normal) AST/SGOT > ULN Version 1, May 12, 2010 Calcium > ULN
14. Inability to sign informed consent
15. Psychological, familial, sociological or geographical conditions which do not permit regular medical follow-up and compliance with the protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-02; Primary Completion 2013-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Toxicity | 24 months

SECONDARY OUTCOMES:
Survival | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Konstantin Lavrenkov, MD, PhD, Principal Investigator — Soroka University Medical Center
Locations (1):
- Soroka University Medical Center, Beersheba, Israel